CLINICAL TRIAL: NCT00424229
Title: Phase II Study of the Efficacy and Safety of Lenalidomide in Adult Subjects With Intermediate-2-or Higt Risk Myelodysplastic Syndrome(MDS) Associated With a Deletion (DEL) 5q [31]
Brief Title: Lenalidomide in Subjects With intermediate2 or High MDS Associated With a Deletion (DEL) 5q [31]
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-REV-2006-02
Record Dates: First submitted 2007-01-15; First posted 2007-01-18 (Estimated); Last update posted 2007-03-12 (Estimated); Status verified 2007-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS INT-2MDS HIGH RISKDELETION 5q[31]Lenalidomide
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: LENALIDOMIDE

SUMMARY:
We are evaluating the incidence of significant hematological response, according to IWG criteria including CR, PR or, major HI, (HI-E, Hl-N,or Hl- P), and cytogenetic response of patients diagnosed with intermediate-2 or high-risk (International Prognostic Scoring System [IPSS]) MDS with a deletion (del) 5q[31]

DETAILED DESCRIPTION:
Subjects meeting all inclusion and exclusion criteria will receive lenalidomide

lenalidomide will be administered at 10 mg (two 5 mg capsules) once daily on Days 1-21, every 4 weeks.

Bone marrow aspirate (baseline and during the course of the study at week 8, 16, 32, 52 and when clinically indicated/for assessment of disease progression) evaluations

Subjects may participate in the study for up to 52 weeks ( in patients still responding after 52 weeks, the drug wil continue to be supplied).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years at the time of signing the informed consent form
* MDS with IPSS scores Int-2 or high with deletion 5q(31)
* Prior thalidomide allowed
* Documented diagnosis of MDS (RA, RARS, RAEB, RAEB-T and CMML with WBC < 13,000/mm3 according to FAB classification) that meets IPSS criteria for intermediate-2 or high-risk disease and has an associated del 5q[31] (the deleted chromosomal region must include 5q[31]), with or without additional cytogenetic abnormalities

Exclusion Criteria:

* Pregnant or lactating females
* Prior therapy with lenalidomide
* MDS with IPSS scores low or Int-1
* Clinical neuropathy of greater than grade 2
* Proliferative (WBC ≥ 13,000/mL) chronic myelomonocytic leukemia (CMML)
* Recombinant human erythropoietin (rHuEPO) therapy received within 28 days
* Use of androgens other than for treating hypogonadism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49
Dates: Start 2006-10; Study Completion 2008-10

PRIMARY OUTCOMES:
Primary: Complete Response; Partial ResponseSecondary: Hematological Improvement

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FENAUX, Profesor, Study Director — Groupe Francophone des Myelodysplasies; Sara Burcheri, Study Director — Groupe français des myélodysplasies
Locations (11):
- France (11):
  - CHU Angers, Angers
  - CHRU Hurriez, Lille
  - Hopital Paoli Calmette, Marseille
  - Hopital Hotel Dieu, Nantes
  - Hopital Archet, Nice
  - Hoiptal St Louis, Paris
  - Hopital Cochin, Paris
  - Hopital Jean-Bernard, Poitiers
  - Centre Henry Becquerel, Rouen
  - Chu Purpan, Toulouse
  - CHU Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Ades L, Boehrer S, Prebet T, Beyne-Rauzy O, Legros L, Ravoet C, Dreyfus F, Stamatoullas A, Chaury MP, Delaunay J, Laurent G, Vey N, Burcheri S, Mbida RM, Hoarau N, Gardin C, Fenaux P. Efficacy and safety of lenalidomide in intermediate-2 or high-risk myelodysplastic syndromes with 5q deletion: results of a phase 2 study. Blood. 2009 Apr 23;113(17):3947-52. doi: 10.1182/blood-2008-08-175778. Epub 2008 Nov 5. PMID 18987358